CLINICAL TRIAL: NCT05632211
Title: A First-in-human, Randomized, Parallel Group, Double-blind, 3-arm Study to Investigate the Comparative PK, Safety, and Tolerability Between Subcutaneous AVT05, US-licensed Simponi®, and EU-approved Simponi® in Healthy Adult Participants
Brief Title: A Study to Investigate the PK, Safety, and Tolerability Between AVT05, US and EU Simponi® in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVT05-GL-P01
Record Dates: First submitted 2022-11-11; First posted 2022-11-30 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinded/unblinded site teams
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AVT05 50mg s.c. (Experimental): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Biological: AVT05
- EU Simponi 50mg s.c. (Active Comparator): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Biological: Simponi
- US Simponi 50mg s.c. (Active Comparator): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Biological: Simponi

INTERVENTIONS:
Biological: AVT05 — Pre filled syringes filled with AVT05
  Arms: AVT05 50mg s.c.
Biological: Simponi — Pre filled syringes filled with Simponi
  Other Names: Golimumab
  Arms: EU Simponi 50mg s.c.; US Simponi 50mg s.c.

SUMMARY:
Rationale:

Alvotech is developing AVT05 globally as a proposed biosimilar to the reference product Simponi (golimumab) for subcutaneous (SC) use. This is a first-in-human (FIH) clinical study with AVT05. The study aims to demonstrate pharmacokinetic (PK) similarity of the proposed biosimilar test product AVT05 and the reference products EU approved Simponi and US-licensed Simponi, in addition to evaluating the safety and tolerability of AVT05, when administered as a single 50 mg/0.5 mL SC dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in the protocol.
* Participants must be 18 to 55 years old (inclusive) at the time of signing the ICF.
* Have a body weight of 50.0 to 90.0 kg (inclusive) and body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive).

Exclusion Criteria:

* Have a history of relevant drug and/or food allergies.
* Known or suspected clinically relevant drug hypersensitivity to golimumab, AVT05, or any of its constituents, which in the opinion of the PI, contraindicates the participant's participation.
* Have any past or concurrent medical conditions that could potentially increase the participant's risks or that would interfere with the study evaluation, procedures, or study completion. Examples of these include medical history with evidence of clinically relevant pathology (eg, malignancies or demyelinating disorders).
* Previous exposure to other TNF-α inhibitors including golimumab.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wynne, Principal Investigator — New Zealand Clinical Research
Locations (2):
- New Zealand Clinical Research, Christchurch, New Zealand
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynne C, Lorch U, Krantz E, Katial R, Ashdown T, Luque M, Sattar A, Rai M, Vashishta L, Petrovic K, Ruffieux R, Leutz S, Berti F. Pharmacokinetic Similarity of Biosimiliar AVT05 Versus Reference Product Golimumab in Healthy Adults: A Double-Blind, Three-Arm, Parallel-Group Study. BioDrugs. 2026 Jan;40(1):121-133. doi: 10.1007/s40259-025-00749-7. Epub 2025 Nov 10. PMID 41212475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVT05 50mg s.c. | EU Simponi 50mg s.c. | US Simponi 50mg s.c.
Started | 115 | 111 | 110
Completed | 112 | 110 | 107
Not Completed | 3 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Other reasons | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVT05 50mg s.c. | EU Simponi 50mg s.c. | US Simponi 50mg s.c. | Total
Number analyzed (Participants) | 115 | 111 | 110 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (8.17) | 29.2 (8.43) | 28.3 (8.16) | 28.6 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 62 | 191
  Male | 50 | 47 | 48 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 17 | 19 | 19 | 55
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 2 | 5
  Black or African American | 43 | 39 | 44 | 126
  White | 46 | 36 | 39 | 121
  More than one race | 1 | 4 | 1 | 6
  Unknown or Not Reported | 5 | 11 | 4 | 20
Weight [Mean (Standard Deviation); unit: kilograms] | 67.74 (9.888) | 67.08 (10.286) | 67.42 (9.736) | 67.42 (9.946)

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate the PK Similarity of AVT05 With US Licensed and EU Approved Simponi and the PK of EU Approved Simponi With US Licensed Simponi
Description: The primary PK parameters to be compared is Cmax and AUC0-inf.
Time Frame: Day zero to day 75 - days 1 (within the hour prior to dosing and at 8 and 12 hours post-dose), 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 22, 29, 36, 43, 50, 57, 64, and 75.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AVT05 50mg s.c. | EU Simponi 50mg s.c. | US Simponi 50mg s.c.
Number analyzed (Participants) | 114 | 111 | 106
ng/mL | 3453.8 (52) | 3468.6 (50) | 3567.1 (51)

2. Primary Outcome: To Demonstrate the PK Similarity of AVT05 With US Licensed and EU Approved Simponi and the PK of EU Approved Simponi With US Licensed Simponi
Description: The primary PK parameter to be compared is AUC0-inf
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | AVT05 50mg s.c. | EU Simponi 50mg s.c. | US Simponi 50mg s.c.
Number analyzed (Participants) | 114 | 111 | 106
ng·h/mL | 1423639 (38) | 1362263 (40) | 1414744 (37)

ADVERSE EVENTS:
Time Frame: From time of signing the ICF until the end of the participant's participation in the study, , approximately 15 weeks.
Arm/Group | AVT05 50mg s.c. | EU Simponi 50mg s.c. | US Simponi 50mg s.c.
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/111 | 0/110
Serious Adverse Events (participants affected / at risk) | 1/115 | 1/111 | 0/110
Other Adverse Events (participants affected / at risk) | 74/115 | 74/111 | 74/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVT05 50mg s.c. (N=115) | EU Simponi 50mg s.c. (N=111) | US Simponi 50mg s.c. (N=110)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVT05 50mg s.c. (N=115) | EU Simponi 50mg s.c. (N=111) | US Simponi 50mg s.c. (N=110)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 13 (13) | 14 (15)
Influenza (Infections and infestations) | 6 (6) | 5 (6) | 7 (7)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 20 (23) | 13 (14) | 20 (26)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 5 (6) | 4 (4) | 7 (7)
Injection site erythema (General disorders) | 5 (5) | 5 (5) | 4 (4)
Vessel puncture site bruise (General disorders) | 3 (3) | 5 (6) | 5 (5)
Injection site pain (General disorders) | 2 (2) | 6 (9) | 2 (2)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1)
Catheter site related reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Puncture site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 7 (7) | 5 (5) | 3 (3)
Mycobacterium tuberculosis complex test positive (Investigations) | 1 (1) | 4 (4) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 5 (6) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 3 (3)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: part 1 (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT05632211/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: part 2 (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT05632211/Prot_SAP_001.pdf